CLINICAL TRIAL: NCT05573880
Title: The Influence of Whole-body Vibration Training on Postural Stability in People With Generalized Joint Hypermobility
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gdansk University of Physical Education and Sport (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: AWFiS/2022_EP
Record Dates: First submitted 2022-09-14; First posted 2022-10-10 (Actual); Last update posted 2022-10-10 (Actual); Status verified 2022-08

CONDITIONS: Hypermobility, Joint
MeSH Terms: conditions — Joint Instability

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- generalized joint hypermobility (Experimental)
  Interventions: Device: Galileo Med35
- without generalized joint hypermobility (Experimental)
  Interventions: Device: Galileo Med35

INTERVENTIONS:
Device: Galileo Med35 — whole-body vibration training on the platform

SUMMARY:
The aim of this study was the assessment of muscle flexibility after 2-weeks of whole-body vibration (WBV) training in people with generalized joint hypermobility (GJH). The study included 33 participants aged 22-25 years. 12 participants were classified into the GJH group and 21 into the control group (CG). The study included the Beighton score and muscle flexibility tests: straight leg raise test (SLR), popliteal angle test (PA), and the modified Thomas test. These tests were performed before and after the short-term WBV program, which consisted of six sessions (frequency: 15 Hz and 30 Hz, amplitude 3 mm, 3 trials x 3 min.).

ELIGIBILITY:
Inclusion Criteria:

* healthy young adults

Exclusion Criteria:

* rheumatological disease
* orthopaedic disease
* neurological disease
* genetic disease
* cardiovascular system disease
* previous injuries of lower limbs
* surgeries of lower limbs and spine
* pain over 3 months of lower limbs and spine
* pregnancy
* implants
* the benign joint hypermobility syndrome (the Brighton criteria)
* the absence during one or more training day

Ages: 22 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2022-08-22 (Actual); Primary Completion 2022-09-05 (Actual); Study Completion 2022-09-05 (Actual)

PRIMARY OUTCOMES:
Beigthon score | Before the main test of muscles flexibility and whole-body vibration training
  The test consisted of the abduction of the thumb to the forearm, the knee hyperextension above 10 degrees, the extension of the metacarpophalangeal joint in the 5th finger above 90 degrees, the elbow hyperextension above 10 degrees, and the placing flat hands on the floor. Each positive test scored 1 point.

SECONDARY OUTCOMES:
Straight Leg Raise Test | Twice - before and after 2-weeks of the whole-body vibration training
  The participant laid in a supine position. The researcher 1 controlled the position of the participant and raised their lower extremity with the knee extended to the first resistance of the hamstring. The researcher 2 assessed the range of hip flexion with an inclinometer, which was placed 10 cm proximally to the patella.

OTHER OUTCOMES:
Popliteal Angle Test | Twice - before and after 2-weeks of the whole-body vibration training
  The participant laid in a supine position with the hip flexed to 90˚ and the extended untested lower extremity. The researcher 1 controlled this position with a goniometer. In this position, the participant had to straighten his knee. The researcher 2 assessed the popliteal angle with an inclinometer, which was placed 10 cm below the tibial tuberosity
Modified Thomas Test | Twice - before and after 2-weeks of the whole-body vibration training
  The modified Thomas test was used to assess the flexibility of One-JHF and Two-JHF. During One-JHF test, the participant laid in a supine position with the pelvis close to the edge of the table. The untested lower extremity was flexed at the hip and knee joint. The researcher 1 controlled and stabilized the participant's position. The tested lower extremity was placed in a relaxed position behind the table. The researcher 2 assessed the range of hip extension/flexion with the inclinometer, which was placed 10 cm proximally to the patella. During the Two-JHF test, the participant was in the same position. The researcher 1 assessed the range of knee flexion with the inclinometer, which was placed 10 cm below the tibial tuberosity

CONTACTS AND LOCATIONS:
Overall Officials: Paulina W Ewertowska, PhD, Study Chair — Gdansk University of Physical Education and Sport
Locations (1):
- Gdansk University of Physical Education and Sport, Gdansk, Pomeranian Voivodeship, Poland

IPD SHARING:
Plan to Share IPD: No